CLINICAL TRIAL: NCT04990609
Title: A Single-arm Phase II Study to Evaluate the Safety and Efficacy of Combination Systematic Chemotherapy and Multiple Rounds of Endoscopic Ultrasound-guided Radiofrequency Ablation in Pancreatic Cancer
Brief Title: EUS-RFA PANCARDINAL-1 Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nirav C Thosani, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-21-0066; R01CA277161-01A1 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-08-04 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: Endoscopic Ultrasound Radiofrequency ablation (EUS-RFA)
MeSH Terms: interventions — Endosonography; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy (NAC) plus endoscopic ultrasound (EUS) radiofrequency ablation (RFA) (Experimental)
  Interventions: Device: Endoscopic Ultrasound (EUS)-Guided Radiofrequency Ablation (RFA); Drug: Neoadjuvant Chemotherapy (NAC)

INTERVENTIONS:
Device: Endoscopic Ultrasound (EUS)-Guided Radiofrequency Ablation (RFA) — Endoscopic ultrasound (EUS)-guided radiofrequency ablation (RFA) consists of the application of an alternating current with a frequency of 350-500 kilohertz (kHz) to the target tissue via a special electrode located at the tip of an echoendoscope. The alternating current causes the vibratory movement of ionic particles in the abutting and adjoining tissue and results in the generation of heat. However, RFA induces not only local disruption of the tumor by heat, but it also produces localized coagulation necrosis of the tumor; which induces the release of large amounts of cellular debris. This cellular debris represents a source of tumor antigens that can trigger a host adaptive immune response against the tumor.
Drug: Neoadjuvant Chemotherapy (NAC) — The NAC regimen will be determined clinically by the participant's physician [possible regimens are either mFOLFIRINOX or Gemcitabine Nab-Paclitaxel +/- Cisplatin (GemAbraxane)].

SUMMARY:
The objectives of this study are to determine the feasibility, tolerability, and treatment effect of endoscopic ultrasound (EUS) radiofrequency ablation (RFA) plus standard-of-care neoadjuvant chemotherapy (NAC) in the treatment of pancreatic ductal adenocarcinoma (PDAC). Endoscopic ultrasound (EUS) radiofrequency ablation (RFA) and neoadjuvant chemotherapy (NAC) will be performed before tumor resection surgery, with the goal of shrinking a tumor or stopping the spread of cancer so that surgery might be less invasive and more effective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed and histologically-confirmed PDAC by biopsy
* Permanent street address
* Consent to study participation
* Axial CT scan consistent with PDAC
* No prior chemotherapy or less than 2 months of pre-operative chemotherapy for PDAC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* Male or female patients < 18 years of age
* No permanent street address or telephone number
* Pregnant patients
* Inmates or prisoners
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are able to complete neoadjuvant chemotherapy plus EUS-RFA and later undergo surgical tumor resection | From the time of EUS-RFA NAC intervention to the time of surgical tumor resection (about 5-6 months)

SECONDARY OUTCOMES:
Radiographic treatment response as assessed by standard Response evaluation criteria in solid tumors (RECIST) criteria | 2 months after the initiation of chemotherapy
  Using the RECIST criteria, treatment response is categorized as follows:
  * Complete response (CR): Disappearance of all target lesions
  * Partial response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
  * Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
  * Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Radiographic treatment response as assessed by standard Response evaluation criteria in solid tumors (RECIST) criteria | 4 months after the initiation of chemotherapy
  Using the RECIST criteria, treatment response is categorized as follows:
  * Complete response (CR): Disappearance of all target lesions
  * Partial response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD
  * Stable disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
  * Progressive disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Number of participants with post-operative complications | from the time of surgical tumor resection to 90 days following surgical tumor resection
Disease-free survival time | from the time of diagnosis to time of recurrence (or up to 5 years after diagnosis, whichever occurs first)
  Disease is defined as clinical evidence of local or distant recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Thosani, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No